CLINICAL TRIAL: NCT03196388
Title: Enzalutamide and External Beam Hypofractionated Radiotherapy For Intermediate Risk Localized Prostate Cancer
Acronym: ENZART
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Canaria de Investigación Sanitaria (Other)
Collaborators: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-004617-25
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Prostate Carcinoma
Keywords: ENZALUTAMIDE; External Beam Hypofractionated Radiotherapy Intermediate Risk Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enzalutamide with External (Experimental): On this study patients will be treated with 6 months of Xtandi (enzalutamide). Approximately one-third of the way through this treatment they will receive EBRT. Starting on Day 1, all patients will ingestenzalutamide 160 mg/day at the same time each day without breaks (except as outlined for toxicity), with or without food, for 6 (28 day +/-3 days) cycles. Dose reduction of enzalutamide to 120 mg/day is allowed with the approval of the Medical Monitor. Patients will be instructed to return all unused capsules at each study visit to assess compliance and will receive study drug every 28 days (+/-3 days) for 6 cycles (25 weeks).
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Radiation: External Beam Radiation Dose will be normalized such that exactly 98% of the PTV (planned target volume) receives the prescription dose and will be scored as per protocol. The maximum allowable dose within the PTV is 107% of the prescribed dose to a volume that is at least 0.03 cc. The minimum allowable dose within the PTV is >95% of the prescribed dose to a volume that is at least 0.03 cc.
  EBRT shall receive prescription doses to the PTV 70 Gy delivered in 2.5 Gy
  Other Names: XTANDI

SUMMARY:
This research study is evaluating a drug called enzalutamide in combination with external beam radiation therapy as a possible treatment for prostate cancer. Presently, when participants receive hormonal therapy with radiation therapy for prostate cancer, medications are given to reduce testosterone levels in the blood stream. This leads to side effects such as loss of sex drive, erectile dysfunction (ED) and decrease in muscle strength. The purpose of this study is test another form of hormonal therapy with radiationtherapy. The medication called enzalutamide will be used with radiation therapy. Instead of lowering testosterone, enzalutamide blocks testosterone in cells. This study will test if enzalutamide when used with radiation will lower the PSA without causing the side effects associated with medications that lower testosterone in the blood stream

DETAILED DESCRIPTION:
The participant will be given a study drug-dosing diary for each of 6 treatment cycles. Each treatment cycle lasts 28 days (4 weeks), during which time the participant will be taking the study drug enzalutamide by mouth (4 pills daily). The diary will also include special instructions for taking the enzalutamide.

The participant will also be undergoing external beam radiation therapy during the study, for a duration of 5,5 weeks. Treatment will be administered on an outpatient basis. This part of the study is considered standard of care.

The participant will be required to have IGRT either by ConeBeam CT study and/or fiducial markers placed within the prostate as part of this study. These are very small gold markers that are placed in the prostate. This procedure is similar to the biopsy that the participant had to diagnose their cancer. These both procedures are routinely performed to permit imaging and position corrections to improve the precision of the external beam (radiation) delivery (Image Guided Radiation Therapy). This is also considered standard of care and is not experimental.

Planned Follow-up: Participants will be followed on study at a 3 month follow-up after treatment (cessation of enzalutamide). Additional follow-up to assess the status of the participant's cancer will be conducted at the discretion of the treating physicians as part of the participant's routine medical care.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of greater than 1 year.
* Diagnosis of histologically confirmed prostate carcinoma
* ECOG Score ≤ 1
* Participants must have an adequate organic function, defined as:

  1. Leukocytes ≥3,000/mcL
  2. Platelets ≥80,000/mcL
  3. Total bilirubin < 2X institutional upper limit
  4. AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  5. Creatinine < 2x institutional limits .
* Potentially fertile patients should use effective contraceptive methods (barrier methods plus other contraceptive methods) before entering the study and during their participation in the study
* Ability to understand and the willingness to sign a written informed consent
* Patients should be available for clinical follow-up.
* To be able to swallow the medication of the study and to fulfill the requirements of the same one

Exclusion Criteria:

* Received an investigational agent within 4 weeks prior to enrollment
* Stage T4 prostate cancer by clinical examination or radiologic evaluation.
* Hypogonadism or severe androgen deficiency as defined by screening serum testosterone less than 50 ng/dL below the normal range for the institution.
* Prior androgen deprivation, chemotherapy, surgery, or radiation for prostate cancer.
* Receiving concurrent androgens, anti-androgens, estrogens, or progestational agents, or received any of these agents within the 6 months prior to enrollment or having taken finasteride or dutasteride within 30 days of registration.
* History of another active malignancy within the previous 5 years other than curatively treated nonmelanomatous skin cancer and superficial bladder cancer. Participants treated for malignancy with no relapse within two years are eligible to participate in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection. Severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrollment.
* History of seizure or any condition or concurrent medication that may predispose to seizure.
* History of loss of consciousness or transient ischemic attack within 12 months prior to enrollment.
* Clinically significant cardiovascular disease, including:

  1. Myocardial infarction within 6 months of enrollment
  2. Uncontrolled angina within 3 months of enrollment
  3. Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multi-gated acquisition scan performed within 3 months results in a left ventricular ejection fraction ≥ 45%;
  4. History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes);
  5. History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
  6. Hypotension as indicated by systolic blood pressure < 86 mmHg on 2 consecutive measurements at the Screening visit;
  7. Bradycardia as indicated by a heart rate < 50 beats per minute at the Screening visit;
  8. Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg on 2 consecutive measurements at the screening visit;
  9. EKG demonstrating equal to or greater than grade III toxicity according the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
* History of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of oral study drug(s) within 3 months of enrollment.
* Major surgery within 4 weeks of registration.
* Previous use, or participation in a clinical trial, of an investigational agent that blocks androgen synthesis (e.g., abiraterone acetate, TAK-700, TAK-683, TAK-448) or targets the androgen receptor (e.g., enzalutamide, BMS 641988); ketoconazole.
* Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, places the patient at undue risk, or complicates the interpretation of safety data.
* Use of herbal or alternative remedies that may affect hormonal status such as Prostasol or PC-SPES.

Ages: 18 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with more or equal 80% reduction of baseline PSA | 25 week after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Carlos Lara Jiménez, MD, PhD, Principal Investigator — Hospital Universitario de Gran Canaria Dr. Negrín
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain

REFERENCES:
- [Result] Boccon-Gibod L, Tombal B. Open to debate. The motion: Hormonal blockade should be limited due to significant adverse effects. Eur Urol. 2009 Jan;55(1):240-3. doi: 10.1016/j.eururo.2008.10.006. Epub 2008 Oct 14. No abstract available. PMID 18930581
- [Result] Keating NL, O'Malley AJ, Freedland SJ, Smith MR. Diabetes and cardiovascular disease during androgen deprivation therapy: observational study of veterans with prostate cancer. J Natl Cancer Inst. 2010 Jan 6;102(1):39-46. doi: 10.1093/jnci/djp404. Epub 2009 Dec 7. PMID 19996060
- [Result] Taylor LG, Canfield SE, Du XL. Review of major adverse effects of androgen-deprivation therapy in men with prostate cancer. Cancer. 2009 Jun 1;115(11):2388-99. doi: 10.1002/cncr.24283. PMID 19399748
- [Result] Tyrrell CJ, Kaisary AV, Iversen P, Anderson JB, Baert L, Tammela T, Chamberlain M, Webster A, Blackledge G. A randomised comparison of 'Casodex' (bicalutamide) 150 mg monotherapy versus castration in the treatment of metastatic and locally advanced prostate cancer. Eur Urol. 1998;33(5):447-56. doi: 10.1159/000019634. PMID 9643663
- [Result] Tran C, Ouk S, Clegg NJ, Chen Y, Watson PA, Arora V, Wongvipat J, Smith-Jones PM, Yoo D, Kwon A, Wasielewska T, Welsbie D, Chen CD, Higano CS, Beer TM, Hung DT, Scher HI, Jung ME, Sawyers CL. Development of a second-generation antiandrogen for treatment of advanced prostate cancer. Science. 2009 May 8;324(5928):787-90. doi: 10.1126/science.1168175. Epub 2009 Apr 9. PMID 19359544
- [Result] Belikov S, Oberg C, Jaaskelainen T, Rahkama V, Palvimo JJ, Wrange O. FoxA1 corrupts the antiandrogenic effect of bicalutamide but only weakly attenuates the effect of MDV3100 (Enzalutamide). Mol Cell Endocrinol. 2013 Jan 5;365(1):95-107. doi: 10.1016/j.mce.2012.10.002. Epub 2012 Oct 11. PMID 23063623
- [Result] Scher HI, Fizazi K, Saad F, Taplin ME, Sternberg CN, Miller K, de Wit R, Mulders P, Chi KN, Shore ND, Armstrong AJ, Flaig TW, Flechon A, Mainwaring P, Fleming M, Hainsworth JD, Hirmand M, Selby B, Seely L, de Bono JS; AFFIRM Investigators. Increased survival with enzalutamide in prostate cancer after chemotherapy. N Engl J Med. 2012 Sep 27;367(13):1187-97. doi: 10.1056/NEJMoa1207506. Epub 2012 Aug 15. PMID 22894553
- [Result] Trump D. Commentary on: "Enzalutamide monotherapy in hormone-naive prostate cancer: primary analysis of an open-label, single-arm, phase 2 study." Tombal B, Borre M, Rathenborg P, Werbrouck P, Van Poppel H, Heidenreich A, Iversen P, Braeckman J, Heracek J, Baskin-Bey E, Ouatas T, Perabo F, Phung D, Hirmand M, Smith MR. Institut de Recherche Clinique, Universite Catholique de Louvain, Brussels, Belgium. Electronic address: bertrand.tombal@uclouvain.be. Aarhus University Hospital, Aarhus, Denmark. Herlev Hospital, Herlev, Denmark. AZ Groeninge Kortrijk, Kortrijk, Belgium. UZ Leuven, Leuven, Belgium. Klinik und Poliklinik fur Urologie, RWTH University Aachen, Aachen, Germany. Rigshospitalet, University of Copenhagen, Copenhagen, Denmark. UZ Brussel, Brussels, Belgium. Univerzita Karlova v Praze, Prague, Czech Republic. Astellas Pharma Global Development, Leiden, Netherlands. Astellas Pharma Global Development, Northbrook, IL, USA. Medivation Inc, San Francisco, CA, USA. Massachusetts General Hospital Cancer Center, Boston, MA, USA: Lancet Oncol. 2014 May;15(6):592-600; doi: 10.1016/S1470-2045(14)70129-9. [Epub 2014 Apr 14]. Urol Oncol. 2016 May;34(5):248-9. doi: 10.1016/j.urolonc.2015.03.012. Epub 2015 Apr 30. PMID 25937426
- [Result] Tombal B, Borre M, Rathenborg P, Werbrouck P, Van Poppel H, Heidenreich A, Iversen P, Braeckman J, Heracek J, Baskin-Bey E, Ouatas T, Perabo F, Phung D, Baron B, Hirmand M, Smith MR. Long-term Efficacy and Safety of Enzalutamide Monotherapy in Hormone-naive Prostate Cancer: 1- and 2-Year Open-label Follow-up Results. Eur Urol. 2015 Nov;68(5):787-94. doi: 10.1016/j.eururo.2015.01.027. Epub 2015 Feb 14. PMID 25687533
- [Result] Fizazi K, Scher HI, Miller K, Basch E, Sternberg CN, Cella D, Forer D, Hirmand M, de Bono JS. Effect of enzalutamide on time to first skeletal-related event, pain, and quality of life in men with castration-resistant prostate cancer: results from the randomised, phase 3 AFFIRM trial. Lancet Oncol. 2014 Sep;15(10):1147-56. doi: 10.1016/S1470-2045(14)70303-1. Epub 2014 Aug 4. PMID 25104109
- [Result] Loriot Y, Miller K, Sternberg CN, Fizazi K, De Bono JS, Chowdhury S, Higano CS, Noonberg S, Holmstrom S, Mansbach H, Perabo FG, Phung D, Ivanescu C, Skaltsa K, Beer TM, Tombal B. Effect of enzalutamide on health-related quality of life, pain, and skeletal-related events in asymptomatic and minimally symptomatic, chemotherapy-naive patients with metastatic castration-resistant prostate cancer (PREVAIL): results from a randomised, phase 3 trial. Lancet Oncol. 2015 May;16(5):509-21. doi: 10.1016/S1470-2045(15)70113-0. Epub 2015 Apr 14. PMID 25888263
- See also: Cross-sectional study of bone turnover during bicalutamide monotherapy for prostate cancer — http://dx.doi.org/10.1016/S0090-4295(02)02006-X